CLINICAL TRIAL: NCT06204055
Title: The Derivation of a Clinical Prediction Rule to Identify Those With Low Back Pain Who Will
Brief Title: The Derivation of a Clinical Prediction Rule to Identify Those With Low Back Pain Who Will Respond Favorably to Intramuscular Dry-needling
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Whitworth University (Other)
Responsible Party: Principal Investigator, Dominic Severino, Assistant Professor, Whitworth University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 878_Severino
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Dry-Needling; Myofascial Pain; Treatment Based Classification
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: The first phase will be an RCT, 2 x 3 group (IMDN or Sham) by time (pretest, post-treatment week 1, post-treatment week 2, posttest, follow-up) with repeated measures on timeframe.
  The second phase will utilize logistic regression analysis to identify associations between the groups' demographic, historical, clinical variables and short-term pain and disability outcomes. This type of analysis will be able to identify strong predictors of the treatment outcome. Various processes will be used to determine optimal model fit for analysis.
Who Masked: Participant
Masking Description: After the physical examination has been performed, each participant will be randomized to receive IMDN or SIMDN. Randomization will be completed by use of a computer-generated list of random numbers that will designate group assignment. The PI will inform the study PTs of the participants group assignment. The list will be maintained by a research assistant who is not involved with participant recruitment, examination or treatment. Participants will be blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intramuscular Dry-Needling (Experimental): (IMDN) is a minimally invasive procedure where a solid filament needle is inserted into a myofascial trigger point.
  Interventions: Other: Intramuscular Dry-Needling
- Sham Intramuscular Dry-Needling (Sham Comparator): ). Park sham acupuncture needles (AcuPrime) will be used to perform sham needling for this group. The sham needle functions by allowing the blunted needle to cause a pricking sensation when pushed against the skin, but does not penetrate. This will allow the patient to perceive that the needle is entering the skin while also maintaining therapist-patient contact and interaction time
  Interventions: Other: Intramuscular Dry-Needling

INTERVENTIONS:
Other: Intramuscular Dry-Needling — It is a minimally invasive procedure where a solid filament needle is inserted deeply into a myofascial trigger point (MTrP) within a muscle in an attempt to abate it and illicit a desired treatment effect.

SUMMARY:
The purpose of this study is to investigate specific clinical characteristics, amongst those with low back pain, that identify patient appropriateness for Intermuscular Dry-Needling (IMDN) and to develop a prediction tool that can be used by clinicians.

DETAILED DESCRIPTION:
The aim of the CPR is to identify patients with LBP who are likely to benefit from IMDN. Improvement of patient-reported outcomes and clinical measures of pain are the outcomes being predicted by the model. The CPR will be developed in a double-phase design. The first phase will be an RCT, 2 x 3 group (IMDN or Sham) by time (pretest, post-treatment week 1, post-treatment week 2, posttest, follow-up) with repeated measures on timeframe. This design will establish if improvement of patient reported outcomes and clinical measures of pain are achieved because of the IMDN treatment. Furthermore, each group will receive the same type and volume of lumbar and hip stretching exercises in conjunction with their assigned needling regimen. The second phase will utilize logistic regression analysis to identify associations between the groups' demographic, historical, clinical variables and short-term pain and disability outcomes. This type of analysis will be able to identify strong predictors of the treatment outcome. Various processes will be used to determine optimal model fit for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 18 and 60 years with non-traumatic low back pain between the 12th rib and the buttock region.
* Participants must also report an Oswestry Disability Index score of at least 20/100 points.

Exclusion Criteria:

* Participants must be able to speak and read English.
* Individuals who are currently pregnant, currently taking pain narcotic medication or have had a prior surgery in the lumbosacral spine
* Those participants whose BMI is greater than 35

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index | Baseline, week 1, week 2 and week 3
  self reported questionnaire that is used to measure a patient's permanent functional disability.

SECONDARY OUTCOMES:
Fear-Avoidance Beliefs Questionnaire | Baseline, week 1, week 2 and week 3
  self reported questionnaire that is used to measure a patient's fear associated with movement and/or work
11 point Numeric Pain-Rating Scale | Baseline, week 1, week 2 and week 3
  self reported scale that is used to rate subjective intensity of back and leg pain

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Severino, PT,DPT, Principal Investigator — Whitworth University
Locations (1):
- Whitworth University, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No